CLINICAL TRIAL: NCT03771989
Title: Treatment of Osteoarthritis With Autologous, Microfragmented Adipose Tissue. A Randomized Controlled Trial
Brief Title: Treatment of Osteoarthritis With Autologous, Microfragmented Adipose Tissue.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kristoffer Barfod, Associate Professor, MD PhD, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TOMAT
Record Dates: First submitted 2018-12-09; First posted 2018-12-11 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study is performed as a blinded, multicenter, randomized, controlled trial with participants individually randomized to one of two parallel groups:
  1. The intervention group: Participants receive one intra articular injection with autologous, microfragmented adipose tissue.
  2. The control group: Participants receive one intra articular injection with Saline (placebo).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: 4.4.1 Randomization Randomization is computer based, performed in blocks of twelve.
  4.4.2 Blinding Blinding of the patient is secured as follows: The liposuction and microfragmentation of the fatty tissue is performed in the operating theatre. When the graft is ready for use the randomization envelope is opened by the project nurse; if the patient is allocated to active treatment syringes containing the microfragmented fatty tissue are prepared; if the patient is allocated to placebo syringes containing saline are prepared. The 10ml syringe is placed in the hand of the treating surgeon. Injection is performed with a 21G cannula. Due to the difference in viscosity of the graft and saline, the surgeon cannot be blinded.
  In order to investigate if the blinding is working the patients will be asked at 6 months follow up which group he/she believe he/she was assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Patients are treated with an intra articular injection with autologous, micro-fragmented adipose tissue.
  Interventions: Biological: autologous, micro-fragmented adipose tissue
- Control (Placebo Comparator): Patients are treated with an intra articular injection with saline (placebo).
  Interventions: Other: Saline

INTERVENTIONS:
Biological: autologous, micro-fragmented adipose tissue — The active treatment is an intra-articular injection with autologous, microfragmented adipose tissue prepared using the Lipogems system.
  Implantation of the graft is performed with the patient supine using two injections sites in order to reduce the risk of extra-articular injection.
  Arms: Intervention
Other: Saline — The placebo is an injection with saline
  Arms: Control

SUMMARY:
The study is a blinded, multicenter, randomized, controlled trial with participants individually randomized to one of two parallel groups:

1. The intervention group: Participants receive one intra articular injection with autologous, microfragmented adipose tissue.
2. The control group: Participants receive one intra articular injection with Saline (placebo).

The objective of the study is to investigate if intra-articular injection with autologous, microfragmented adipose tissue prepared using the Lipogems system affects the patient reported outcome in patients with osteoarthritis of the knee.

The primary endpoint is KOOS4 evaluated at 6 months after the intervention. Secondary endpoints are the KOOS including all five subscales evaluated after 6months, 1 and 2 years.

DETAILED DESCRIPTION:
2 Study Objective To investigate if intra-articular injection with autologous, microfragmented adipose tissue prepared using the Lipogems system affects the patient reported outcome in patients with osteoarthritis of the knee.

Hypothesis Treatment with autologous, microfragmented adipose tissue has the potential to reverse degenerative changes in knees with osteoarthritis. The patient will experience a better patient reported health in comparison with placebo treatment.

Null hypothesis There is no difference in patient reported outcome when treatment with autologous, microfragmented adipose tissue is compared to placebo treatment.

3 Background Osteoarthritis (OA) of the knee is a destructive joint disease, causing degeneration of cartilage, damage to the underlying bone and morphological changes to the joint1. It is a major public health concern due to the increased life expectancy of the ageing population2,3. No approved medical treatment that reverses the morphological changes currently exists. Conventional treatment includes physiotherapy, pain killers, braces and in end-stage OA surgical knee replacement4.

During the past decade researchers have started to explore the regenerative potential of mesenchymal stem cells (MSC) in OA5. MSCs are multipotent progenitor cells able to give rise to osteocytes, adipocytes, chondrocytes, myoblasts and tenocytes6. MSCs were first used to treat Chondral defects in 19987 and to treat OA in 20028. Since then, a number of case reports and prospective series have been published showing significant short term and long term effect on pain and cartilage thickness5. Latest a prospective case-series of 1128 patients involving 1856 joints showed an improvement of at least 50% in 86% of patients at 3 months and 91% of patients at 12 months using a modified Knee/Hip Osteoarthritis Outcome Score (KOOS/HOOS) questionnaire9. Only 0.9% of patients did not show improvement after treatment. However, when interpreting these studies one should bear in mind that they are all level four evidence and as such prone to bias.

No serious adverse effects like infection or neoplastic formation have been observed in treatment with MSC of OA9,10. Non-manipulated or minimally manipulated cell therapies have been used within a wide range of medical conditions including: stroke, myocardial infarction, Crohn's disease, rheumatoid arthritis and breast augmentation. More than 17.000 scientific articles have been published reporting treatment of more than 320.000 patients11. No severe safety issues have been raised12.

Mesenchymal stem cells can be derived from bone marrow or adipose tissue5. Most research has been performed on bone marrow-derived stem cells. Studies have shown promising results, but in 2016 a randomized study found no effect of active treatment with bone marrow aspirate concentrate compared to placebo with saline in the treatment of arthritic knees13. The past years a series of studies have been published showing promising effect of Adipose-derived mesenchymal stem cells (AMSCs). By using AMSC a large amount of cells can be harvested from a small volume of tissue thereby avoiding the costly and time consuming process of expanding the cells in culture5,9.

Mesenchymal stem cells are thought to be able to activate and influence the microenvironment by serving as "a site-regulated drug store" 14. The use of adipose-derived mesenchymal stem cells in treatment of OA has had a huge interest the past years15,16, and the complex regulatory issues applying for enzymatic treated and/or expanded cells have led to the development of minimally manipulated tissue17. The Lipogems system is one such system where the adipose tissue is microfragmented and washed free of blood residues. The resulting product is safe (FDA approval in 2016) and is said to be effective in the treatment of different pathologies18, but level one evidence is lacking.

In a pilot study of 20 patients with knee OA performed by the research group behind the present project the Lipogems system showed promising results (submitted). No safety issues were raised and the patients improved from 13 to 21 in the five sub scales of KOOS at 3 and 12 months follow up. The Lipogems system is introduced at the Danish market in 2018. There is a pressing need to perform a state of the art RCT comparing the Lipogems system with placebo in the treatment of knee OA.

4 Design of the study 4.1 Patient involvement in the study design In order to secure the highest degree of relevance of the study qualitative interviews were conducted with 10 patients suffering from OA of the knee who would be considered eligible for inclusion. They were asked the following two questions: 1) What is your biggest problem in concern to your knee(s)? 2) What are your most important criteria of success after a procedure to your knee(s)? Based on the answers endpoints were developed and chosen.

4.5 Time schedule Inclusion of patients is planned to begin 15th of November 2018. The expected study period is 4 years; the recruitment itself is expected to span 1½ year, provided that an average of 8 patients is included per month.

4.6 Termination of the trial If a critical adverse event is considered to have a causal relationship with the treatment the project manager is responsible to initiate a discussion with the other investigators on whether the trial should be terminated.

4.7 Follow up Follow up investigations are performed after 3, 6, 12 and 24 months. Study nurse 1 performs follow up in the outpatient clinic. If patients do not show for follow up investigation they will be contacted by phone up to three times and will be asked to return fulfilled questionnaires by mail.

4.8 Data registration All relevant data is recorded RedCap in a database specifically designed for the trial. The data registration will be reported to the Danish Data Protection Agency.

The following data is registered:

4.8.1 Inclusion Date of examination. Social security number Demographic parameters: Age, gender. Risk parameters: ASA score, smoking, diabetes, coronary heart disease, rheumatic disease (RA or connective tissue disease).

Type of work Sports activity KOOS Tegner Activity Scale Kellgren-Lawrence score

4.8.2 Follow up at 3, 6 and 12 months Date of examination. Change in work status Sports activity KOOS Tegner Activity Scale Donor site morbidity

4.9 Biological material

A research biobank is created for storage of tissue. The following tissue will be stored:

Samle of the graft.

5 Population Patients who are suffering from pain and functional impairment due to osteoarthritis of the knee and referred to one of the participating departments are eligible for inclusion. Patients who fulfil the inclusion criteria but do not wish to participate are treated according the standard regimen of the department.

5.1 Inclusion procedure Patients referred to the orthopaedic department at the involved hospitals are seen in the outpatient clinic. If they fulfil the inclusion criteria they will be verbally informed of the study, given written patient information, and offered an appointment with study nurse 1 and an investigating surgeon.

At this appointment it is re-assessed whether the patient meets the inclusion criteria. If so the patient will once again be verbally informed of the study and given the opportunity - on informed basis without any pressure - to decide whether he/she wants to participate in the trial. The patient is informed of his/her right to 24 hours of reflection.

All patients assessed for eligibility are registered according to the consort requirements.

7 Safety 7.1 Risks and side effects The project team has performed a pilot study raising no major safety issues (the resulting manuscript is submitted for publication). Non-manipulated or minimally manipulated cell therapies have been used within a wide range of medical conditions including: stroke, myocardial infarction, Crohn's disease, rheumatoid arthritis and breast augmentation. More than 17,000 scientific articles have been published reporting treatment of more than 320,000 patients11. No severe safety issues have been raised12. However, there is always the risk of unknown side effects.

7.2 Education and training Trained personnel at the investigation sites will carry out treatment, observations and measurements.

7.3 Adverse events In this context adverse events are defined as any unintended, unfavourable finding, symptom or disease that occurs, whether it is considered to be related to the study or not. Adverse events will be recorded.

8 Statistics 8.1 Sample Size 120 patients will be included; 60 patients in each group. The sample size calculation is based on a clinical relevant difference of 10 point in KOOS, a standard deviation (SD) of 15 and power of 0.90 (two sided). 98 patients are required; due to the risk of drop out 120 patients will be included; 60 in each group. The used SD and clinical relevant difference are recommended at KOOS.NU

. 8.2 Analysis of endpoints The two groups are described descriptively regarding demographic parameters as well as primary and secondary endpoints. Comparison of the primary and secondary outcomes of both groups is done by use of relevant statistics according to the characteristics and distribution of the variables. The change of the outcomes over a period of time is described within each group.

All statistical testing will be performed at the two-sided 5% significance level, and 95% confidence intervals will be presented where appropriate. No formal interim analyses are planned, and hence no statistical testing will take place until the one-year analysis. The one year analysis will take place after all participants have completed their one year follow-up and sufficient time has been allowed for data entry and validation.

Prior to any analysis, missing data pattern will be investigated and reasons for missing data obtained and summarized where possible. The primary analysis will be conducted as an intention-to-treat analysis, which includes all participants with missing outcome data, unless there is clear evidence that its underlying assumption is inappropriate. Sensitivity analysis will be performed to assess the robustness of the results by imputing missing data using multiple imputations under both missing at random and missing not at random assumptions. Per protocol analyses will also be performed.

11 Ethics 11.1 Ethical considerations The study is carried out in accordance with the principles of the Helsinki Declaration.

11.2 Declaration of consent All patients will receive verbal and written information concerning the study. The inclusion will take place after a declaration of consent has been obtained. It is the responsibility of the investigators to provide patients with comprehensive verbal and written information concerning the course of the study, purpose, potential risks and benefits.

12 Data processing All Data will be stored in RedCap. The patients will be identified by an assigned number. At the completion of the study all identifiable data will be destroyed. The project will be reported to the Danish Data Protection Agency. The project will follow the Danish act concerning storage and handling of personal data.

ELIGIBILITY:
5.2 Inclusion criteria

* Age 18-70 years.
* Kellgren-Lawrence grade 2 - 3 in the tibiofemoral joint
* The patient must be expected to be able to attend follow up examinations
* The patient must be able to speak and understand Danish
* The patient must be able to give informed consent

5.3 Exclusion criteria

* Smoking (the patient must consent to being non-smoking 6 weeks pre and post the procedure)
* Varus or valgus malalignment of the knee > 5 degrees
* Laxity of the MCL or LCL of 10 degrees or more compared to the opposite knee
* Knee instability and anterior-posterior laxity of 3mm or above
* Preceding open surgery to the knee or fracture in the proximal tibia or distal femur
* Extension deficit of the knee
* Kellgren-Lawrence grade 4 in any of the three compartments
* BMI > 40
* Terminal illness or severe medical illness: ASA score higher than or equal to 3

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
KOOS4 | 6 months
  The Knee injury and Osteoarthritis Outcome Score. The KOOS questionnaire was developed in the 1990s as an instrument to assess the patient's opinion about their knee and associated problems. Since the first publication in 1998, the psychometric properties of the KOOS have been assessed in more than twenty individual studies from all over the world. Furthermore, KOOS has been evaluated and compared to other instruments in several reviews measured after one year19,20 ,21,22.
  KOOS4 constructs an average score for four out of the five KOOS subscale scores. It was first used by Frobell et al in 201023. The reason for not including all five subscale scores is that in active patients, very few difficulties with activities of daily living (ADL) exists. Including the subscale ADL would then add unwanted 'noise' to the constructed outcome22.

SECONDARY OUTCOMES:
KOOS | 6 months
  The Knee injury and Osteoarthritis Outcome Score (including all five subscales) The KOOS holds 42 items in five separately scored subscales: KOOS Pain, KOOS Symptoms, Function in daily living (KOOS ADL), Function in Sport and Recreation (KOOS Sport/Rec), and knee-related Quality of Life (KOOS QOL)22,24.
  The five patient-relevant subscales of KOOS are scored separately: KOOS Pain (9 items); KOOS Symptoms (7 items); KOOS ADL (17 items); KOOS Sport/Rec (5 items); KOOS QOL (4 items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as is common in orthopedic assessment scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved22.
KOOS | 12 months
  The Knee injury and Osteoarthritis Outcome Score (including all five subscales) The KOOS holds 42 items in five separately scored subscales: KOOS Pain, KOOS Symptoms, Function in daily living (KOOS ADL), Function in Sport and Recreation (KOOS Sport/Rec), and knee-related Quality of Life (KOOS QOL)22,24.
  The five patient-relevant subscales of KOOS are scored separately: KOOS Pain (9 items); KOOS Symptoms (7 items); KOOS ADL (17 items); KOOS Sport/Rec (5 items); KOOS QOL (4 items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as is common in orthopedic assessment scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved22.
KOOS | 24 months
  The Knee injury and Osteoarthritis Outcome Score (including all five subscales) The KOOS holds 42 items in five separately scored subscales: KOOS Pain, KOOS Symptoms, Function in daily living (KOOS ADL), Function in Sport and Recreation (KOOS Sport/Rec), and knee-related Quality of Life (KOOS QOL)22,24.
  The five patient-relevant subscales of KOOS are scored separately: KOOS Pain (9 items); KOOS Symptoms (7 items); KOOS ADL (17 items); KOOS Sport/Rec (5 items); KOOS QOL (4 items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as is common in orthopedic assessment scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved22.
Failure | 6 months
  If the patients do not experience a clinically relevant improvement in KOOS4 the treatment is considered a failure. A clinical relevant difference is estimated to be 10points (please see section 8 Statistics). The number of patients experiencing failure of the treatment is recorded at each follow up.
Failure | 12 months
  If the patients do not experience a clinically relevant improvement in KOOS4 the treatment is considered a failure. A clinical relevant difference is estimated to be 10points (please see section 8 Statistics). The number of patients experiencing failure of the treatment is recorded at each follow up.
Failure | 24 months
  If the patients do not experience a clinically relevant improvement in KOOS4 the treatment is considered a failure. A clinical relevant difference is estimated to be 10points (please see section 8 Statistics). The number of patients experiencing failure of the treatment is recorded at each follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Kristoffer W Barfod, Principal Investigator — Copenhagen University Hospital Hviovre
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Barfod KW, Blond L, Mikkelsen RK, Bagge J, Holmich LR, Kallemose T, Troelsen A, Holmich P. Treatment of knee osteoarthritis with a single injection of autologous micro-fragmented adipose tissue is not superior to a placebo saline injection: a blinded randomised controlled trial with 2-year follow-up. Br J Sports Med. 2025 Aug 26;59(17):1219-1227. doi: 10.1136/bjsports-2024-108732. PMID 40101939